CLINICAL TRIAL: NCT05346913
Title: Internet-Delivered Cognitive Behaviour Therapy Program for Caregivers of Persons With Spinal Cord Injury: A Pilot Study
Brief Title: ICBT Program for Caregivers of Persons With SCI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Swati Mehta, Scientist, Principle Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 118285P2
Record Dates: First submitted 2022-04-21; First posted 2022-04-26 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Internet-Delivered Cognitive Behavioural Therapy; Depression; Anxiety; Spinal Cord Injuries; Caregiver Burnout
MeSH Terms: conditions — Depression; Anxiety Disorders; Spinal Cord Injuries; Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Caregivers of Persons with Spinal Cord Injury (mTBI) (Experimental)
  Interventions: Behavioral: Internet-delivered Cognitive Behavioural Therapy(ICBT)

INTERVENTIONS:
Behavioral: Internet-delivered Cognitive Behavioural Therapy(ICBT) — ICBT provides online structured self-help modules over several months based on the principles of CBT in combination with weekly guidance through emails and telephone calls. The course comprises 6 online lessons that provide psychoeducation about: 1) symptom identification and the cognitive behavioural model; 2) thought monitoring and challenging; 3) de-arousal strategies and pleasant activity scheduling; 4) graduated exposure/pacing; 5) memory and attention; and 6) relapse prevention. Participants will also have the opportunity to ask any questions regarding the content of the program materials and will receive a response from their Guide within 48-72 hours. Guide will spend ~15 mins. per week/per participant. All Guides have completed a university program (psychology or social work) and are registered clinicians or students working under supervision of a registered clinician.

SUMMARY:
Spinal cord injuries have a devastating effect on individuals incurring the life changing event; however, the injury can also affect those who are integrally involved in their care. Assisting individuals after an SCI frequently falls on unpaid, family caregivers. Studies have reported that caregivers experienced significantly greater negative outcomes than positives. The most common negative outcome factors were high levels of burden, poor adjustment to role, decreased QOL, emotional distress, and strain on relationships. Burden of care was also associated with lower levels of functioning of the care recipient, demonstrating the integral relationship between those who provide care and those who receive it. Considering their importance in maintaining their care recipient's wellbeing post-injury, caregivers require ongoing support as a central part of the wider healthcare system. Numerous caregivers are unprepared to handle the responsibilities of their role and lack specialized training to efficiently cope with the burden. Guided internet-delivered CBT (ICBT) offers an accessible and flexible approach for psychosocial service delivery in the community. Evidence for the effectiveness of ICBT has been reported in various populations. The results from our study provide evidence for the potential of guided ICBT to improve psychosocial outcomes among those with SCI. Enhancing the overall wellbeing of the caregiver has previously been shown to improve outcomes of those with SCI. However, evidence for the acceptability and effectiveness of an ICBT approach among caregivers is lacking; as a first step, we plan to conduct a feasibility study of ICBT for SCI caregivers.

ELIGIBILITY:
Inclusion Criteria:

1. adults ≥ 18 years
2. have provided care to a person with SCI in the community for a period of over six months post injury
3. report elevated symptoms of anxiety and/or depression
4. access to a computer and the internet
5. cognitive capacity to read and understand the content of the intervention.

Exclusion Criteria:

1. high risk of suicide
2. primary problems with psychosis, alcohol or drug problems, mania
3. currently receiving active psychological treatment for anxiety or depression
4. concerns about online therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Change in Depression | Time Frame: Baseline to 3 months
  Patient Health Questionnaire - 9 Item (PHQ-9). Higher total scores indicate greater severity of depression. Scores range from 0 to 27.
Change in Caregiver Burden | Time Frame: Baseline to 3 months
  Craig Caregiver Assessment of Reward and Effort. Higher scores indicate greater caregiver. Scores range from 0 to 96.

SECONDARY OUTCOMES:
Change in Anxiety | Time Frame: Baseline to 3 months
  Generalize Anxiety Disorder - 7 Item (GAD7). Higher total scores indicate greater severity of anxiety. Scores range from 0 to 21.
Change in quality of life | Time Frame: Baseline to 3 months
  The Visual Analogue Scale of the EuroQol five-dimension (EQ-5D) questionnaire will be used. Higher numbers indicates poorer quality of life. Scores range from 0 to 100

CONTACTS AND LOCATIONS:
Overall Officials: Swati Mehta, PhD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's